CLINICAL TRIAL: NCT05099861
Title: Clinical Anatomy of Superficial Veins of Lower Limbs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, MUDr. Michaela Hronova, MUDr., Charles University, Czech Republic
Other Study IDs: CHU185797621
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Saphenous Vein Injury
Keywords: small saphenous vein; great saphenous vein; saphenopopliteal junction; venae intersaphenae

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: Healthy volunteers with no sign of internal disease. Age 18-50, both women and men.
  Interventions: Other: No intervention
- patients with internal disease: Patients with internal disease, both women and men.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — this is an observational study

SUMMARY:
The study is focused on clinical anatomy of superficial veins of lower limbs. We are mapping their anatomy via ultrasonography. We are focusing on saphenopopliteal junction and communicants between small saphenous vein and great saphenous vein.

DETAILED DESCRIPTION:
Research project is focused on superficial veins of lower extremities, especially their clinical anatomy. Superficial veins are located within the compartimentum saphenum. The function of superficial veins is drainage of intradermal and epifascial spaces. Superficial veins and their function are fundamental in development of chronic venous disorder. These veins are physiologically connected with deep venous system via perforators but also between each other via communicanting veins. Communicanting veins between small saphenous vein and great saphenous vein have not been described yet, particularly because of their variations. Clinically important is also the saphenopopliteal junction in the fossa poplitea. This region features many variations, which were described in many studies. Also, the nomenclature of saphenopopliteal juction is not standardised in comparison to the saphenofemoral junction. Moreover, many articles are pointing out that there were not specified all potential drainage ways of the cranial extension of small saphenous vein (extesio cranialis). Articles are uniform neither in its prevalence nor in its terminology.

The knowledge of connections between the superficial and deep venous systems as well as knowledge of communicanting veins between superficial veins is important for diagnosis and proper treatment of chronic venous disorder. Variabilities of these veins can play fundamental role in choosing the proper graft for aorto-coronary bypass grafting. The ununiformed nomenclature of superficial veins, their communicating veins and junctions can cause misleading preoperative diagnosis and overlooking of these structures in clinical practise.

ELIGIBILITY:
Inclusion Criteria:

* women and men
* age 18-80

Exclusion Criteria:

* wounds on lower limbs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: European population
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
The Anatomy of superficial Veins of Lower Limbs | 2022-2024
  the anatomy observed by ultrasonography imaging focus on communicans between small saphenous vein and great saphenous vein

SECONDARY OUTCOMES:
The Anatomy of Superficial Veins of Lower Limbs: junction saphenopopliteal | 2022-2024
  clinical anatomy of saphenopopliteal junction and its variations observed by ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Hronová, doctor, Principal Investigator — 1. faculty of Medicine, Charles University
Locations (1):
- First faculty of medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided